CLINICAL TRIAL: NCT05602298
Title: The Validity of the Quality of Recovery Score 15 Following Cardiac Surgery
Brief Title: The Quality of Recovery-15 Survey After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Terri Sun, Clinical Associate Professor, University of British Columbia
Other Study IDs: H22-01459
Record Dates: First submitted 2022-07-11; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Disease; Surgery; Surgery-Complications; Cardiac Valve Disease; Cardiac Complication; Cardiac Event
MeSH Terms: conditions — Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of Recovery 15 survey — QOR 15 is a patient reported outcomes measure (PROM) tool used as a global measure of patient recovery after surgery and anesthesia. It uses fifteen questions to assess various domains of patient health: pain, physical comfort, physical independence, psychological support, and emotional state.

SUMMARY:
Patient reported outcomes are becoming increasingly recognized as an important metric to determine efficacy of interventions following recovery after cardiac surgery. Quality of Recovery 15 survey is a tool that attempts to measure patients' recovery across several different domains (i.e physical, emotional and social). This tool has been validated extensively in the post operative patient population, but these studies contained only small numbers of cardiac surgery patients. This population faces unique challenges to recovery such as a longer duration of mechanical ventilation, ICU and hospital LOS, delirium, significant pain in the first 24-48 hours and post operative arrhythmias. This study aims to validate the QoR 15 in this population exclusively to determine if it is feasible, valid, reliable and responsive in this unique population.

DETAILED DESCRIPTION:
The QoR-15 will be administered at three time points, verbally to the patient by a standardized script. The time points are at baseline QoR-15 (t=0) at time of enrollment in the PAC, surgical daycare or surgical ward, post extubation day 1 (t=2), and post extubation day 2 (t=3) and 12 weeks following surgery. Concurrently, patients will also be asked to rate their overall postoperative recovery using an 100-mm visual analogue scale (VAS), from "poor recovery" to "excellent recovery". A subset of patients will also be asked to repeat the QoR 15 questionnaire 30-60 min later to measure repeatability. Duration to complete each QoR-15 will be recorded.

Baseline demographic information (sex, age, ethnicity, comorbidities such as smoking status, lung disease, history of MI, hypertension, heart failure, renal failure, NYHA class) will be collected at time of enrollment. Intraoperative data (type of surgical procedure, duration of procedure, duration of cardiopulmonary bypass and aortic cross clamp time), Cardiac Surgery Intensive Care Unit (CSICU) LoS, duration of mechanical ventilation, and hospital LoS will be collected following patient discharge from hospital.

Post operative complications will be assessed using the Clavien-Dindo Classification, which is a 5 scale classification system, ranking complications on severity, depending on therapy required. Days alive and at home to Day 30 (DAH 30) (10) is a quantifiable and patient centred outcome that may be used as a proxy for a patient's recovery after surgery. This will be collected from chart review at 30 days following surgery and will be used as a metric to assess construct validity.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing cardiac surgery (outpatient or inpatient surgery)

Exclusion Criteria:

* At baseline patient screening:

  1. Patients who have severe cognitive impairment (score of 1 or 2) measured through the use of the three minute screening tool, Mini-Cog 26
  2. Patient has limited ability to complete assessment at baseline
  3. Unable to read/speak English
  4. Significant hearing impairments
  5. Critical state before surgery with high probability of death within 24 hours
* After cardiac surgery, patients will be removed from further data collection if:

  1. They require a tracheostomy or 5 days of ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing inpatient or outpatient cardiac surgery at St. Paul's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the QoR 15 (1.1) | Aug 4, 2022 to Jan 1, 2023
  Response rate (Percentage of questionnaires completed at each time point)
Feasibility of the QoR 15 (1.2) | Aug 4, 2022 to Jan 1, 2023
  Proportion of questions completed independently without help/clarification by research assistant (Percentage)
Feasibility of the QoR 15 (1.3) | Aug 4, 2022 to Jan 1, 2023
  Proportion of questions completed/answered (Percentage)
Feasibility of the QoR 15 (1.4) | Aug 4, 2022 to Feb 1, 2023
  Time taken to complete the questionnaire (median +/- IQR)
Validity (2.1) | Aug 4, 2022 to Feb 1, 2023
  Correlation between QoR 15 compared with VAS global rating of health using 100mm scale (Pearson correlation coefficient)
Validity (2.2) | Aug 4, 2022 to Feb 1, 2023
  Correlation with NRS pain score (Pearson correlation coefficient)
Validity (2.3) | Aug 4, 2022 to Feb 1, 2023
  Association between QoR 15 with age, gender, duration of surgery, duration of ICU stay, duration of hospital stay, opioid consumption, surgical complications and DAH 30 will be assessed using multivariable linear regression
Reliability (3.1) | Aug 4, 2022 to Feb 1, 2023
  Internal consistency - averaged correlation between each item with QoR15
Reliability (3.2) | Aug 4, 2022 to Feb 1, 2023
  15-25 patients will be asked to repeat a second time 30-60min later and their QoR 15 score compared
Reliability (3.3) | Aug 4, 2022 to Feb 1, 2023
  Inter-item correlation matrix
Reliability (3.4) | July 18. 2022 to Jan 1, 2023
  Interdimensional and item total dimension correlation
Responsiveness (4.1) | July 18. 2022 to Jan 1, 2023
  Cohen effect size (avg change scores from pretest to post tes, divided by SD at baseline Standardised response mean (change scores divided by SD of change scores)

CONTACTS AND LOCATIONS:
Overall Officials: Alana Flexman, Study Director — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Background] Campfort M, Cayla C, Lasocki S, Rineau E, Leger M. Early quality of recovery according to QoR-15 score is associated with one-month postoperative complications after elective surgery. J Clin Anesth. 2022 Jun;78:110638. doi: 10.1016/j.jclinane.2021.110638. Epub 2022 Jan 13. PMID 35033845